CLINICAL TRIAL: NCT01626859
Title: A Pharmacokinetic Study of MP-214 in Patients With Schizophrenia (12 Weeks Treatment Study)
Brief Title: A Pharmacokinetic Study of MP-214 in Patients With Schizophrenia
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Tanabe Pharma Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: A002-A11
Record Dates: First submitted 2012-06-19; First posted 2012-06-25 (Estimated); Results first posted 2021-04-12 (Actual); Last update posted 2026-01-05 (Actual); Status verified 2025-12

CONDITIONS: Schizophrenia
Keywords: Schizophrenia; Antipsychotic Agents; Mental Disorder; Psychotropic Drugs; Dopamine Agents; Central Nervous System Agents
MeSH Terms: conditions — Schizophrenia; Mental Disorders

ARMS (3):
- MP-214 3mg (Experimental)
  Interventions: Drug: MP-214 3mg
- MP-214 6mg (Experimental)
  Interventions: Drug: MP-214 6mg
- MP-214 9mg (Experimental)
  Interventions: Drug: MP-214 9mg

INTERVENTIONS:
Drug: MP-214 3mg — Patients who meet eligibility criteria will be administered a once daily oral 3mg of MP-214 for twelve weeks.
  Arms: MP-214 3mg
Drug: MP-214 6mg — Patients who meet eligibility criteria will be administered a once daily oral 6mg of MP-214 for twelve weeks.
  Arms: MP-214 6mg
Drug: MP-214 9mg — Patients who meet eligibility criteria will be administered a once daily oral 9mg of MP-214 for twelve weeks.
  Arms: MP-214 9mg

SUMMARY:
The objective of this study is to evaluate the pharmacokinetics, safety and efficacy of MP-214 in patients with schizophrenia.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent obtained from the patient before the initiation of any study-specific procedures
* Patients diagnosed with schizophrenia according to the diagnostic criteria of the Diagnostic and Statistical Manual of Mental Disorders, Fourth Edition, Text Revision (DSM-IV-TR) criteria for schizophrenia
* Patients with normal physical examination, laboratory, vital signs, and/or electrocardiogram (ECG)

Exclusion Criteria:

* Patients with a DSM-IV-TR diagnosis of schizoaffective disorder, schizophreniform disorder, other psychotic disorders other than schizophrenia, or bipolar I or II disorder

The information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Ages: 20 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 38 (Actual)
Dates: Start 2012-05; Primary Completion 2013-08 (Actual); Study Completion 2013-08 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Sakai, Osaka, Japan

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | MP-214 3mg | MP-214 6mg | MP-214 9mg
Started | 11 | 16 | 11
Completed | 9 | 8 | 7
Not Completed | 2 | 8 | 4
Not completed — Adverse Event | 1 | 3 | 2
Not completed — Physician Decision | 0 | 1 | 0
Not completed — Withdrawal by Subject | 1 | 4 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | MP-214 3mg | MP-214 6mg | MP-214 9mg | Total
Number analyzed (Participants) | 11 | 16 | 11 | 38
Age, Continuous [Mean (Standard Deviation); unit: years] | 43.2 (13.2) | 43.1 (10.7) | 43.2 (13.3) | 43.1 (11.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 9 | 6 | 20
  Male | 6 | 7 | 5 | 18

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Events as a Measure of Safety and Tolerability
Time Frame: Up to 24 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | MP-214 3mg | MP-214 6mg | MP-214 9mg
Number analyzed (Participants) | 11 | 16 | 11
Participants | 11 | 15 | 11

2. Primary Outcome: Maximum Plasma Concentration of Unchanged MP-214, M7 (Desmethyl Cariprazine) and M6 (Didesmethyl Cariprazine) at Day 84
Time Frame: On Day 84 samples were taken pre-dose and 3, 4, 6 and 8 hours post-dose.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | MP-214 3mg | MP-214 6mg | MP-214 9mg
Number analyzed (Participants) | 11 | 16 | 11
ng/mL
  Unchanged MP-214 | 10.23 (4.691) | 22.65 (4.181) | 28.77 (8.024)
  M7 (desmethyl cariprazine) | 2.624 (1.521) | 5.963 (1.593) | 8.550 (3.750)
  M6 (didesmethyl cariprazine) | 15.77 (10.88) | 35.94 (7.995) | 51.82 (32.71)

3. Primary Outcome: Time to Maximum Plasma Concentration of Unchanged MP-214, M7 (Desmethyl Cariprazine) and M6 (Didesmethyl Cariprazine) at Day 84
Time Frame: On Day 84 samples were taken pre-dose and 3, 4, 6 and 8 hours post-dose.
Measure: Mean (Standard Deviation); unit: hour
Arm/Group | MP-214 3mg | MP-214 6mg | MP-214 9mg
Number analyzed (Participants) | 11 | 16 | 11
hour
  Unchanged MP-214 | 3.31 (0.52) | 3.31 (1.02) | 3.58 (0.60)
  M7 (desmethyl cariprazine) | 4.45 (1.21) | 4.77 (2.14) | 5.60 (1.22)
  M6 (didesmethyl cariprazine) | 7.76 (9.21) | 7.34 (6.83) | 7.56 (7.27)

4. Primary Outcome: Area Under the Plasma Concentration-Time Curve From Time Zero to 24 Hours of Unchanged MP-214, M7 (Desmethyl Cariprazine) and M6 (Didesmethyl Cariprazine) at Day 84
Time Frame: On Day 84 samples were taken pre-dose and 3, 4, 6 and 8 hours post-dose.
Measure: Mean (Standard Deviation); unit: ng*h/mL
Arm/Group | MP-214 3mg | MP-214 6mg | MP-214 9mg
Number analyzed (Participants) | 11 | 16 | 11
ng*h/mL
  Unchanged MP-214 | 155.96 (71.99) | 358.37 (85.24) | 466.36 (154.55)
  M7 (desmethyl cariprazine) | 50.03 (31.19) | 115.26 (23.47) | 163.31 (72.72)
  M6 (didesmethyl cariprazine) | 352.03 (252.78) | 800.21 (206.73) | 1140.42 (711.59)

ADVERSE EVENTS:
Arm/Group | MP-214 3mg | MP-214 6mg | MP-214 9mg
Serious Adverse Events (participants affected / at risk) | 0/11 | 2/16 | 0/11
Other Adverse Events (participants affected / at risk) | 11/11 | 15/16 | 11/11
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | MP-214 3mg (N=11) | MP-214 6mg (N=16) | MP-214 9mg (N=11)
Schizophrenia (Psychiatric disorders) | 0 | 2 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | MP-214 3mg (N=11) | MP-214 6mg (N=16) | MP-214 9mg (N=11)
Sinus tachycardia (Cardiac disorders) | 0 | 0 | 1
Hyperprolactinaemia (Endocrine disorders) | 1 | 0 | 0
Abnormal sensation in eye (Eye disorders) | 0 | 1 | 0
Cataract (Eye disorders) | 0 | 1 | 0
Conjunctivitis (Eye disorders) | 0 | 1 | 0
Abdominal discomfort (Gastrointestinal disorders) | 0 | 0 | 1
Abdominal distension (Gastrointestinal disorders) | 0 | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 1
Abdominal pain upper (Gastrointestinal disorders) | 1 | 0 | 0
Abdominal tenderness (Gastrointestinal disorders) | 0 | 0 | 1
Constipation (Gastrointestinal disorders) | 0 | 2 | 1
Dental caries (Gastrointestinal disorders) | 1 | 1 | 1
Diarrhoea (Gastrointestinal disorders) | 1 | 1 | 0
Faeces hard (Gastrointestinal disorders) | 0 | 0 | 1
Gastritis (Gastrointestinal disorders) | 2 | 0 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 1 | 0
Haematochezia (Gastrointestinal disorders) | 1 | 0 | 0
Irritable bowel syndrome (Gastrointestinal disorders) | 1 | 0 | 0
Mucous stools (Gastrointestinal disorders) | 0 | 0 | 1
Nausea (Gastrointestinal disorders) | 2 | 1 | 0
Paraesthesia oral (Gastrointestinal disorders) | 0 | 0 | 1
Salivary hypersecretion (Gastrointestinal disorders) | 0 | 0 | 1
Vomiting (Gastrointestinal disorders) | 1 | 2 | 2
Chest discomfort (General disorders) | 0 | 1 | 0
Chills (General disorders) | 0 | 1 | 0
Feeling abnormal (General disorders) | 1 | 0 | 1
Irritability (General disorders) | 0 | 0 | 1
Malaise (General disorders) | 1 | 0 | 0
Pyrexia (General disorders) | 1 | 0 | 0
Hepatic function abnormal (Hepatobiliary disorders) | 0 | 0 | 1
Seasonal allergy (Immune system disorders) | 1 | 0 | 0
Enteritis infectious (Infections and infestations) | 0 | 1 | 0
Gastroenteritis (Infections and infestations) | 0 | 3 | 1
Hordeolum (Infections and infestations) | 0 | 1 | 0
Nasopharyngitis (Infections and infestations) | 3 | 6 | 1
Pulpitis dental (Infections and infestations) | 0 | 1 | 0
Tinea infection (Infections and infestations) | 1 | 0 | 0
Contusion (Injury, poisoning and procedural complications) | 0 | 0 | 1
Excoriation (Injury, poisoning and procedural complications) | 1 | 0 | 0
Laceration (Injury, poisoning and procedural complications) | 0 | 1 | 0
Ligament sprain (Injury, poisoning and procedural complications) | 1 | 0 | 0
Thermal burn (Injury, poisoning and procedural complications) | 1 | 0 | 0
Tooth fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Alanine aminotransferase increased (Investigations) | 1 | 2 | 0
Aspartate aminotransferase increased (Investigations) | 0 | 2 | 0
Blood cholesterol increased (Investigations) | 0 | 1 | 0
Blood creatine phosphokinase increased (Investigations) | 1 | 2 | 0
Blood lactate dehydrogenase increased (Investigations) | 0 | 1 | 0
Blood prolactin increased (Investigations) | 1 | 0 | 1
Blood triglycerides increased (Investigations) | 0 | 1 | 0
Blood uric acid increased (Investigations) | 1 | 0 | 0
Blood urine present (Investigations) | 1 | 0 | 0
Gamma-glutamyltransferase increased (Investigations) | 1 | 0 | 0
Heart rate increased (Investigations) | 1 | 0 | 0
Liver function test abnormal (Investigations) | 0 | 0 | 1
Red blood cell count increased (Investigations) | 0 | 0 | 1
Thyroxine free increased (Investigations) | 0 | 1 | 0
Weight decreased (Investigations) | 1 | 0 | 0
White blood cell count increased (Investigations) | 1 | 2 | 0
Dyslipidaemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Electrolyte depletion (Metabolism and nutrition disorders) | 1 | 0 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Metabolic disorder (Metabolism and nutrition disorders) | 0 | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1
Akathisia (Nervous system disorders) | 5 | 3 | 3
Athetosis (Nervous system disorders) | 0 | 1 | 0
Dizziness (Nervous system disorders) | 0 | 0 | 1
Dizziness postural (Nervous system disorders) | 1 | 0 | 0
Dyskinesia (Nervous system disorders) | 1 | 0 | 0
Extrapyramidal disorder (Nervous system disorders) | 0 | 1 | 0
Facial spasm (Nervous system disorders) | 0 | 1 | 0
Headache (Nervous system disorders) | 1 | 0 | 0
Restless legs syndrome (Nervous system disorders) | 0 | 0 | 1
Sedation (Nervous system disorders) | 0 | 1 | 0
Somnolence (Nervous system disorders) | 0 | 3 | 1
Tremor (Nervous system disorders) | 0 | 3 | 0
Hallucination, visual (Psychiatric disorders) | 0 | 1 | 0
Insomnia (Psychiatric disorders) | 2 | 4 | 3
Restlessness (Psychiatric disorders) | 6 | 4 | 2
Schizophrenia (Psychiatric disorders) | 1 | 5 | 1
Suicidal ideation (Psychiatric disorders) | 1 | 0 | 0
Urinary retention (Renal and urinary disorders) | 0 | 1 | 0
Upper respiratory tract inflammation (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Cold sweat (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Haemorrhage subcutaneous (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Hyperkeratosis (Skin and subcutaneous tissue disorders) | 1 | 1 | 0
Ingrowing nail (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Seborrhoeic dermatitis (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Skin erosion (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Hot flush (Vascular disorders) | 0 | 1 | 0
Hypertension (Vascular disorders) | 1 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other